CLINICAL TRIAL: NCT03366714
Title: Comparison of Efficacy of Noninvasive Ventilation With RAM Cannula Versus Short Bi-nasal Cannula in Respiratory Distress Syndrome of Preterm Infants
Brief Title: RAM Cannula Versus Short Bi-nasal Cannula in Respiratory Distress Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, İsmail Kürşad Gökce, Departman of Pediatrics, Division of Neonatoloji, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017/40
Record Dates: First submitted 2017-11-24; First posted 2017-12-08 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: Noninvasive ventilation, respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RAM cannula (Experimental): nasal CPAP support with RAM cannula
  Interventions: Device: nasal CPAP support with RAM cannula
- Hudson cannula (short binasal cannula) (Active Comparator): nasal CPAP support with Hudson cannula
  Interventions: Device: nasal CPAP support with Hudson cannula

INTERVENTIONS:
Device: nasal CPAP support with RAM cannula — Patients with respiratory distress syndrome who do not need intubation in the delivery room. This groub will be provided with non-invasive respiratory support RAM cannula.
  Arms: RAM cannula
Device: nasal CPAP support with Hudson cannula — Patients with respiratory distress syndrome who do not need intubation in the delivery room. This groub will be provided with non-invasive respiratory support Hudson cannula.
  Arms: Hudson cannula (short binasal cannula)

SUMMARY:
Noninvasive ventilation defines methods of providing ventilation support with constant or variable pressure using nasal or nasopharyngeal interfaces without endotracheal intubation or tracheostomy. Today, short binasal prongs and different types of nasal masks are the most commonly used nasal interfaces in the NICU with the aim of providing NIV.

RAM cannula (Neotech ™, Valencia, CA), a new nasal interface, is increasingly used in NID applications in newborn infants. The RAM cannula is available in the inspiration and expiration arms of the stroke while reducing the dead space in the respiratory tract due to the low nasal prong diameter. There are not enough studies comparing the effectiveness of the RAM cannula with other short binasal prongs or nasal masks.

Investigators compared the effectiveness and nasal injury rates of RAM cannula and short binasal prong as NIV interfaces in preterm infants.

DETAILED DESCRIPTION:
In the past years endotracheal intubation and mechanical ventilation with surfactant therapy was the standard treatment of moderate to severe respiratory distress syndrome (RDS). Especially in the last 10 years, prolonged intubation and positive pressure ventilation have been shown to increase the frequency of bronchopulmonary dysplasia, a kind of chronic pulmonary disease. Intubation and positive pressure ventilation cause volu-trauma, baro-trauma, and alveolar secondary to bio-trauma, leading to excessive distension and inflammation, disrupting alveolar formation, resulting in fibrosis and bronchopulmonary dysplasia. Intubation and mechanical ventilation also involve ventilator-associated pneumonia. For this reason, strategies for lung protective ventilation have become increasingly widespread in recent years and noninvasive ventilation (NNV) applications without endotracheal intubation have become the first choice in neonatal ventilation.

Noninvasive ventilation defines methods of providing ventilation support with constant or variable pressure using nasal or nasopharyngeal interfaces without endotracheal intubation or tracheostomy. Noninvasive ventilation can be performed in a variety of forms such as continuous positive airway pressure (NCPAP) nasal intermittent positive-pressure ventilation (NIPPV) and high-flow nasal cannulae.

Different nasal interfaces are used to provide noninvasive ventilation support. For this purpose, there is no standard apparatus used in neonatal intensive care units (NICU). Nasopharyngeal cannulae are not currently recommended for use with NIV because they cause extensive resistance during spontaneous breathing, nasopharyngeal area damage and colonization, although they have been widely used in previous years. Today, short binasal prongs and different types of nasal masks are the most commonly used nasal interfaces in the NICU with the aim of providing NIV. Nasal interfaces are recommended to be placed on the surface without causing pressure loss. For this purpose, hoods and fixing apparatus are frequently used. For this reason, babies often become restless and agitated during NIV applications. In addition, necrosis and deformities may develop in septum due to pressure of nasal septum.

RAM cannula (Neotech ™, Valencia, CA), a new nasal interface, is increasingly used in NID applications in newborn infants. RAM seems ideal to allow effective and cranium development in the prevention of pressure damage to the face due to the design of the cannula and the need for head or face access to detect it. The RAM cannula is available in the inspiration and expiration arms of the stroke while reducing the dead space in the respiratory tract due to the low nasal prong diameter. Although the use of RAM cannula as a NIV interface in newborn intensive care units is becoming increasingly widespread, the number of studies related to RAM cannula is limited. Most of the studies investigating the effectiveness of this interface were made on artificial lung models. In the study of "Mukerji" and colleagues, the short binasal prong and RAM cannula were compared as interfaces in NIPPV application in the artificial lung model and it was found that carbon dioxide excretion in short binasal prongs was better than RAM cannula with an increase in peak inspiratory pressure. Studies conducted by Iyer and colleagues in the artificial lung model show that RAM leakage rates below 30% lead to adequate pressure transfer to the cannulae, while leakage rates above 50% reduce pressure transfer to the lungs. Similar results have also been found in the work of "Gerdes" et al. A number of studies have been conducted on the clinical use of RAM as a noninvasive ventilation interface and in these studies it has been shown that the use of RAM cannula as an interface in NCPAP, NIPPV or even nasal high frequency ventilation applications to provide NIV is not well tolerated and does not cause gastric perforation or nasal septum damage. In the study of "Nzegwu" et al. It has been shown that in two-thirds of the patients who were treated with RAM cannula and NIV support, the respiratory support was successfully cut off. Nevertheless, none of these studies compared the RAM cannula activity with the other binasal prongs or nasal masks. Investigators compared the effectiveness (rates of surfactant therapy application, rates of intubation, total NIV duration) and nasal injury rates of RAM cannula and short binasal prong as NIV interfaces in preterm infants at neonatal intensive care unit.

Considering the studies made in the artificial lung models of RAM cannulas, which are becoming increasingly widespread in the NICUs, because of their simple and simple design and easy connection to the standard circuits of the ventilators without any intervention, investigators think that the effectiveness of NIV application is insufficient compared to the short binasal cannula.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 26-34 weeks and,
* born in our hospital and,
* Patients with clinical findings (tachypnea, groaning, chest retractions) of RDS

Exclusion Criteria:

* Patients who needed intubation to stabilize in the delivery room or who had severe congenital anomalies.

Ages: 1 Minute to 15 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Nasal IPPV failure | up to four weeks
  Non invasive ventilation failure in patients who underwent nasal IPPV with RAM cannula

SECONDARY OUTCOMES:
NİV duration | up to two months
  In patients with NİV (nasal IPPV) who underwent RAM cannula or short binasal cannula (prong). We compared the time of NIV

CONTACTS AND LOCATIONS:
Locations (1):
- Turgut Özal Medical Center, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis P, Davies M, Faber B. A randomised controlled trial of two methods of delivering nasal continuous positive airway pressure after extubation to infants weighing less than 1000 g: binasal (Hudson) versus single nasal prongs. Arch Dis Child Fetal Neonatal Ed. 2001 Sep;85(2):F82-5. doi: 10.1136/fn.85.2.f82. PMID 11517198
- [Background] Gerdes JS, Sivieri EM, Abbasi S. Factors influencing delivered mean airway pressure during nasal CPAP with the RAM cannula. Pediatr Pulmonol. 2016 Jan;51(1):60-9. doi: 10.1002/ppul.23197. Epub 2015 Apr 7. PMID 25851534
- [Result] Nzegwu NI, Mack T, DellaVentura R, Dunphy L, Koval N, Levit O, Bhandari V. Systematic use of the RAM nasal cannula in the Yale-New Haven Children's Hospital Neonatal Intensive Care Unit: a quality improvement project. J Matern Fetal Neonatal Med. 2015 Apr;28(6):718-21. doi: 10.3109/14767058.2014.929659. Epub 2014 Jun 30. PMID 24874561